CLINICAL TRIAL: NCT06489392
Title: Pterygium Colli Classification of Mehri Turki Imen
Brief Title: Mehri Turki Webbed Neck Classification
Status: Completed | Type: Observational
Sponsor: Mohamed Tahar Maamouri University Hospital (Other)
Responsible Party: Principal Investigator, Imen Turki Mehri, MD, Principal investigator, Mohamed Tahar Maamouri University Hospital
Other Study IDs: Mehri Turki I
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Turner Syndrome; Pterygium Colli; Web Neck; Klippel-Feil Syndrome
Keywords: Webbed neck; Classification; Surgical technique
MeSH Terms: conditions — Turner Syndrome; Klippel-Feil Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to identify all types of congenital neck deformities called " webbed neck ". Through a literature survey, the researcher selected 27 articles describing the surgical treatment of the webbed neck, but without considering the varieties of this deformity. For this reason, the researcher studied all the reported cases from which she developed a classification containing 4 types of webbed necks allowing the use of the most suitable technique to enhance the surgical outcomes.

DETAILED DESCRIPTION:
Through a literature survey of 27 selected articles (from PubMed database and clarivate web of science). The publication years ranged from 1937 to 2020 and the number of patients reported to have undergone surgery was 78 patients.

The webbed neck is a noticeable congenital deformity mainly observed in Turner syndrome. It consists of a bilateral fold extending from the mastoid to the acromion with several distinctions as described in Mehri Turki's webbed neck classification as follows:

Type 1: The fold is maintained by a fibrotic band and the posterior skin is abnormally hairy with a low hairline placement.

Type 2: There is no fibrotic band and the hair abnormality exists as in Type 1

Type 3: There is a fibrotic band and a low posterior hairline but the posterior skin is hairless

Type 4: The fold is maintained by a fibrotic band without hair abnormality

It appears that according to the type of webbed neck, the surgical approach and surgical steps and technique will be adapted to what will be corrected. This classification is therefore crucial to guide surgeons towards the most suitable technique allowing the best results.

ELIGIBILITY:
Inclusion Criteria:

* Articles with a detailed description of the surgical technique
* Articles reporting post-operative results
* Articles written in English or French

Exclusion Criteria:

* Articles with incomplete descriptions of the webbed neck
* Articles without iconography

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study is about 78 patients reported in the literature, aged between 2 and 30 years and born with a webbed neck (or pterygium colli)
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Mehri Turki Webbed neck classification | Baseline, pre-sugical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Imen Mehri Turki, Principal Investigator — Mohamed Tahar Maamouri University Hospital, Nabeul Tunisia
Locations (1):
- Mohamed Tahar Maamouri University hospital, Nabeul, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Data are available in the published article: https://doi.org/10.1007/s10006-023-01166-2

REFERENCES:
- See also: Mehri Turki (2023) Surgical techniques for the webbed neck: a narrative review with a comparative study and surgical decision-making algorithm for an optimal aesthetic result — https://doi.org/10.1007/s10006-023-01166-2